CLINICAL TRIAL: NCT03073564
Title: Effect of Expiratory Positive Airway Pressure on Dynamic Hyperinflation and Ability to Exercise With Upper Limbs in COPD Patients
Brief Title: Effect of Expiratory Positive Pressure on Dynamic Hyperinflation and Ability to Exercise With Upper Limbs in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Dannuey Machado Cardoso, Prof., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-0422
Record Dates: First submitted 2017-02-16; First posted 2017-03-08 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Dyspnea; Cardiopulmonary Exercise Test; Positive-Pressure Respiration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: The first arm of the study consists of the identification of patients who present dynamic hyperinflation (HD) through the incremental cardiopulmonary test for upper limbs. Following the HDP patients will perform a resistance test for the upper limbs with an application of EPAP. A final stage of the study will be a test for the upper limbs with an EPAP application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Incremental cardiopulmonary test (No Intervention): Incremental cardiopulmonary test for upper limbs will be performed only to identify patients who exhibit dynamic hyperinflation during upper limb exercise.
- Endurance test (Experimental): The endurance test for upper limbs will be performed in two conditions: In the first the patients perform the test in usual breathing, without the use of EPAP. In the second the test will be performed using the EPAP mask.
  Interventions: Diagnostic Test: Endurance test for upper limbs
- Functional test (Experimental): The functional test for upper limbs will be performed from protocol already published for the 6-min pegboard and ring test (6PBRT). In this stage the patients will perform the 6PBRT in usual breathing and as the use of the EPAP mask.
  Interventions: Diagnostic Test: Functional test

INTERVENTIONS:
Diagnostic Test: Endurance test for upper limbs — Subjects will initially perform maximal incremental cardiopulmnar test of upper limbs to assess the suggestion of dynamic hyperinflation (DH). After that, it will be randomized, for those who presented DH, to perform the endurance test with and without the use of positive expiratory pressure mask.
  Arms: Endurance test
Diagnostic Test: Functional test — The 6-min pegboard and ring test (6PBRT) will be performed under usual breathing and during application of the EPAP mask. In this condition will be evaluated the presence of dynamic hyperinflation, perception of effort and dipnea, in addition to exercise capacity.
  Arms: Functional test

SUMMARY:
The study will evaluate the effect of positive airway expiratory pressure (EPAP) on patients with chronic obstructive pulmonary disease (COPD) during submaximal upper limb exercise.

DETAILED DESCRIPTION:
The study to be developed from this project aims to evaluate the effect of positive airway expiratory pressure (EPAP) on upper limb exercise-induced dynamic hyperinflation (DH) in patients with chronic obstructive pulmonary disease (COPD). To this end, a cross-over study will be implemented, developed at the Pulmonology Department of Hospital de Clínicas de Porto Alegre. Patients with moderate to very severe, clinically stable COPD will be evaluated. The anthropometric data and pulmonary function will be collected from the medical records, being the study divided into two stages. First stage: At the first visit, dyspnea, quality of life will be evaluated and a maximal incremental cardiopulmonary exercise test (CPET) for upper limb with DH evaluation during exercise. Patients who presented DH on incremental CPET will be invited to return for a second and third visit. In the second and third visit an endurance test will be performed with 80% of the load reached in the incremental CPET and DH determination, one of the tests performed during the application of EPAP through a face mask with pressure level Of 10 cmH2O and another in usual breathing, with the mask without the use of the positive pressure generating valve. The sequence of the test, ie, with and without EPAP, will be obtained through electronic randomization. Patients completing stage 1 will be invited to enter step 2. In this step, which will occur in a single visit, patients will perform a 6-minute pegboard and ring test (6PBRT) with The same monitoring of CPET in three different situations, according to randomization: habitual breathing, half-closed lip breathing (RLS) and the EPAP mask. Thus, it is expected that the application of EPAP through face mask and the use of RLS will reduce DH during submaximal exercise with upper limb, which will be associated with the reduction of dyspnea and increased tolerance to exercise in COPD patients .

ELIGIBILITY:
Inclusion Criteria:

* clinical disease stability (no signs of exacerbation within 8 weeks prior to enrollment)
* receiving standard long-term bronchodilator (BD) therapy
* able to perform cycle ergometer exercise for upper limbs

Exclusion Criteria:

* use artificial airways
* severe comorbidities, such as heart, orthopedic or neurological diseases that are risky or make it impossible to exercise
* Patients on oxygen or with indication of continuous home oxygen therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Dynamic hyperinflation | The inspiratory capacity is assessed at rest before the cardiopulmonary exercise test (CPET) is performed, every two minutes during and immediately after the end of the test. The estimated time of the test will be 8 to 12 minutes.
  Dynamic hypersensitivity is assessed through changes in inspiratory capacity.

SECONDARY OUTCOMES:
Dyspnea | Dyspnea will be evaluated at rest before the cardiopulmonary exercise test (CPET) is performed, every two minutes during and immediately after the end of the test. The estimated time of the test will be 8 to 12 minutes.
  Dyspnea will be assessed by the Borg dispenia perception scale.
Perception of exertion in upper limbs. | Perception of exertion in upper limbs will be evaluated at rest before the cardiopulmonary exercise test (CPET) is performed, every two minutes during and immediately after the end of the test. The estimated time of the test will be 8 to 12 minutes.
  Perforation of exertion in the upper limbs will be assessed through the Borg perception scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marli M Knorst, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vestbo J, Prescott E, Lange P. Association of chronic mucus hypersecretion with FEV1 decline and chronic obstructive pulmonary disease morbidity. Copenhagen City Heart Study Group. Am J Respir Crit Care Med. 1996 May;153(5):1530-5. doi: 10.1164/ajrccm.153.5.8630597.
- [Background] O'Donnell DE, Laveneziana P. Dyspnea and activity limitation in COPD: mechanical factors. COPD. 2007 Sep;4(3):225-36. doi: 10.1080/15412550701480455. PMID 17729066
- [Background] O'Donnell DE, Parker CM. COPD exacerbations . 3: Pathophysiology. Thorax. 2006 Apr;61(4):354-61. doi: 10.1136/thx.2005.041830. PMID 16565268
- [Background] O'Donnell DE, Laveneziana P, Ora J, Webb KA, Lam YM, Ofir D. Evaluation of acute bronchodilator reversibility in patients with symptoms of GOLD stage I COPD. Thorax. 2009 Mar;64(3):216-23. doi: 10.1136/thx.2008.103598. Epub 2008 Dec 3. PMID 19052054
- [Background] Porto EF, Castro AA, Velloso M, Nascimento O, Dal Maso F, Jardim JR. Exercises using the upper limbs hyperinflate COPD patients more than exercises using the lower limbs at the same metabolic demand. Monaldi Arch Chest Dis. 2009 Mar;71(1):21-6. doi: 10.4081/monaldi.2009.372. PMID 19522161
- [Background] Velloso M, Stella SG, Cendon S, Silva AC, Jardim JR. Metabolic and ventilatory parameters of four activities of daily living accomplished with arms in COPD patients. Chest. 2003 Apr;123(4):1047-53. doi: 10.1378/chest.123.4.1047. PMID 12684292
- [Background] Colucci M, Cortopassi F, Porto E, Castro A, Colucci E, Iamonti VC, Souza G, Nascimento O, Jardim JR. Upper limb exercises using varied workloads and their association with dynamic hyperinflation in patients with COPD. Chest. 2010 Jul;138(1):39-46. doi: 10.1378/chest.09-2878. Epub 2010 Mar 4. PMID 20202941
- [Background] Wibmer T, Rudiger S, Heitner C, Kropf-Sanchen C, Blanta I, Stoiber KM, Rottbauer W, Schumann C. Effects of nasal positive expiratory pressure on dynamic hyperinflation and 6-minute walk test in patients with COPD. Respir Care. 2014 May;59(5):699-708. doi: 10.4187/respcare.02668. Epub 2013 Oct 29. PMID 24170913
- [Background] Monteiro MB, Berton DC, Moreira MA, Menna-Barreto SS, Teixeira PJ. Effects of expiratory positive airway pressure on dynamic hyperinflation during exercise in patients with COPD. Respir Care. 2012 Sep;57(9):1405-12. doi: 10.4187/respcare.01481. Epub 2012 Feb 17. PMID 22348429
- [Background] Padkao T, Boonsawat W, Jones CU. Conical-PEP is safe, reduces lung hyperinflation and contributes to improved exercise endurance in patients with COPD: a randomised cross-over trial. J Physiother. 2010;56(1):33-9. doi: 10.1016/s1836-9553(10)70052-7. PMID 20500135
- [Background] van der Schans CP, de Jong W, de Vries G, Kaan WA, Postma DS, Koeter GH, van der Mark TW. Effects of positive expiratory pressure breathing during exercise in patients with COPD. Chest. 1994 Mar;105(3):782-9. doi: 10.1378/chest.105.3.782. PMID 8131541
- [Background] O'Donnell DE, Revill SM, Webb KA. Dynamic hyperinflation and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):770-7. doi: 10.1164/ajrccm.164.5.2012122. PMID 11549531